CLINICAL TRIAL: NCT04432337
Title: Role of Type 2 Diabetes in Potentiating the Inflammatory Response Post Extracorporeal Circulation, Mediated by the NLRP3 Inflammasome, in Patients After Cardiac Surgery
Brief Title: Role of Type 2 Diabetes in Potentiating the Inflammatory Response Post Extracorporeal Circulation After Cardiac Surgery
Acronym: DT2CEC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Departure of the principal investigator
Sponsor: University Hospital Center of Martinique (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 19_RIPH2-15
Record Dates: First submitted 2020-06-11; First posted 2020-06-16 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Inflammatory Response; Extracorporeal Circulation; Complications; Cardiac Surgery; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Type 2 diabetics patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Type 2 diabetes patients (Experimental): The variation in the plasma concentration of the two pro-inflammatory cytokines IL-1β and IL18, between a baseline level measured the day before the operating room (D-1) and 24 hours (D1) for TD2 patients after cardiac surgery with extracorporeal circulation .
  Interventions: Procedure: The role of the activation of the NLRP3 inflammasome after cardiac surgery
- Non-diabetic type 2 patients (Active Comparator): The variation in the plasma concentration of the two pro-inflammatory cytokines IL-1β and IL18, between a baseline level measured the day before the operating room (D-1) and 24 hours (D1) for non-diabetic type 2 patients after cardiac surgery with extracorporeal circulation
  Interventions: Procedure: The role of the activation of the NLRP3 inflammasome after cardiac surgery

INTERVENTIONS:
Procedure: The role of the activation of the NLRP3 inflammasome after cardiac surgery — Determine the effect on the inflammatory response post extracorporeal circulation mediated by the NLRP3 inflammasome, in patients after cardiac surgery

SUMMARY:
Adult cardiac surgery ensures the surgical treatment of valvular and coronary pathologies and of heart failure with the placement of ventricular assistance. Extracorporeal circulation (ECC) is one of the major technical advances associated with cardiac surgery to replace cardiac and pulmonary functions during surgery. ECC can nevertheless lead to postoperative complications, the origin of which is linked to the patient's initial contact with the circuit and membranes of the ECC. This contact triggers a series of humoral and cellular reactions that occur in the first few hours after the ECC and the inflammatory syndrome post ECC fades on its own and usually disappears between the 4th and 6th postoperative day. If the inflammatory response post ECC is most often transient, certain conditions will maintain and intensify this response at the origin of postoperative complications, possibly leading to the patient's death. Among these situations, the investigators find the notion of emergency cardiac surgery, a patient's age over 75 years and a preoperative history of decompensated heart failure, renal failure or type 2 diabetes (T2D).

The inflammasome family of receptors of the nucleotide oligomerization domain (NOD) type, pyrin domain containing 3, NLRP3, is a multi-protein platform of recent discovery which plays a major role in the signaling pathways of the innate inflammatory response.

The role of the activation of the NLRP3 inflammasome in cardiovascular pathologies is now well established and its metabolic priming by hyperglycemia could explain the greater seriousness of these pathologies in T2D patients due to an exacerbated inflammatory response.

What is the effect of T2D status on the inflammatory response post ECC, mediated by the NLRP3 inflammasome, in patients after cardiac surgery?

DETAILED DESCRIPTION:
Adult cardiac surgery provides surgical treatment of valvular, coronary, and heart failure pathologies with the installation of ventricular assistance. Extracorporeal circulation (ECC) is one of the major technical advances associated with cardiac surgery to replace cardiac and pulmonary functions during surgery. However, ECC can lead to postoperative complications, the origin of which is linked to the patient's initial contact with the circuit and membranes of the ECC. This contact triggers a series of humoral and cellular reactions such as activation of the plasma contact system and complement, coagulation and fibrinolysis, activation of endothelial cells and leukocytes, as well as the release into the circulating blood of many mediators of inflammation such as cytokines TNF-α, interleukin IL -1β, interleukin IL6 and interleukin IL8. These reactions occur in the first hours after the ECC and the inflammatory syndrome post ECC fades by itself and usually disappears between the 4th and 6th postoperative day. Different technical and pharmacological modalities (biocompatibility of circuits, hemofiltration, leukocyte filter, antioxidants, anti-inflammatories, corticoids) have helped reduce the inflammatory syndrome post ECC, but their partial effectiveness highlights the need to better understand the molecular mechanisms of inflammation. post ECC in order to improve its prevention.

If the inflammatory response post ECC is most often transient, certain conditions will maintain and intensify this response at the origin of postoperative complications, possibly leading to the patient's death. Among these situations, The investigators find the notion of emergency cardiac surgery, a patient's age> 75 years and a preoperative history of decompensated heart failure, renal failure or type 2 diabetes (T2D).

Defined according to the criteria proposed by the World Health Organization (WHO) and the American Diabetes Association (ADA), DT2 is a major independent risk factor for morbidity and mortality from general surgery, and from surgery especially the heart. The risk of cardiovascular and infectious complications after cardiac surgery in T2D patients increases by 17% for each unit of glycemia above 6 mmol / L. Strict control of blood sugar during the perioperative phase, however, significantly reduces the risk of complications in T2D patients. Physiopathologically, the higher incidence of postoperative complications in T2D patients is attributed to the exacerbation of the postoperative inflammatory response and its deleterious effects on vascular function. A recent study confirms that the expression of messenger RNAs coding for the inflammation genes (IL-1β, IL8) and the transitional activation factors (MYC / JUN) is increased in T2D patients and that this chronic state of low grade preoperative would promote deregulation of the inflammatory response after cardiac surgery, and the occurrence of cardiovascular complications. The level of inflammation in T2D patients is also usually reflected by an increase in plasma levels of proteins in the acute phase of inflammation (C-reactive protein CRP, in particular) and other pro-inflammatory cytokines (TNF-α IL6). These different results suggest that the activation of the NOD-like receptor family pyrin domain containing 3, (NLRP3) inflammasome may play a central role in low-level chronic inflammatory status in T2D patients.

The inflammasome NOD-like receptor family pyrin domain containing 3, NLRP3, is a multi-protein platform whose activation is involved in the signaling pathways of the innate inflammatory response in many inflammatory and infectious diseases, as well as metabolic pathologies like gout and type 2 diabetes. The assembly of the NLRP3 inflammasome results in the activation of inflammatory caspases allowing the cleavage of the pro-cytokines IL-1β and IL-18 into mature and active cytokines. Several studies show that T2D hyperglycemia is a pre-activation or priming factor for NLRP3 which potentiates the secondary activation of NLRP3 and the synthesis of the interleukins of IL-1β and IL18. During T2D, other metabolic signals such as the accumulation of free fatty acids, the release of cellular debris (damage-associated molecular patterns, DAMPs), and reactive oxygen species (ROS) are also responsible for the priming of NLRP3. Among the molecular motifs DAMPs, mitochondrial DNA (mtDNA) is a powerful activator of the NLRP3 inflammasome due to the ancestral bacterial origin of mitochondria.

The role of the activation of the NLRP3 inflammasome in cardiovascular pathologies is now well established and its metabolic priming by hyperglycemia could explain the greater seriousness of these pathologies in T2D patients due to an exacerbated inflammatory response. Currently, there is no human data on the role of NLRP3 inflammasome activation in post-ECC inflammatory syndrome. The investigators envision that the extracorporeal circulation (ECC), responsible for cellular damage, is accompanied by a release of molecular patterns of DAMPs type at the origin of the activation of the NLRP3 inflammasome.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 75 years old
* Type 2 diabetic patients (WHO definition and American Diabetes Association) according to the following criteria: fasting blood glucose ≥ 7.0 mmol / L (fasting = no caloric proportion for at least 8 h) or glycosylated hemoglobin level HbA1c ≥ 6, 5% (in adults), or blood sugar 2 hours after ingestion of 75 g of glucose ≥ 11.1 mmol / L, or random blood sugar ≥ 11.1 mmol / L, either at any time of the day, without seeing at the time of the last meal.
* Patients undergoing aortocoronary bypass surgery or valve replacement with extracorporeal circulation at the university hospital of Martinique
* Patients able to receive and understand information related to research and blood samples taken during treatment
* Patients able to freely express informed and written consent
* Patients supported by french social security

Exclusion Criteria:

* Vulnerable people: people deprived of their liberty by a judicial or administrative decision, subjects admitted to a health or social protection establishment, major subjects under legal protection (guardianship or curatorship) or under the protection of justice, patients in situation emergency. Pregnant or lactating women, or women of childbearing potential without effective contraception. People with a state of health incompatible with the follow-up of the protocol (psychiatric disorders, uncontrolled disease), having cognitive disorders which do not allow the understanding of the study.
* Type 1 diabetic patient
* Patient who has a systemic inflammatory disease
* Patient who has an autoimmune disease
* Patient who has a cancer pathology
* Patient who has contraindications related to surgical operations in general such as general anesthesia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Variation in the plasma concentration of cytokines IL-1β and IL18 | 48 hours
  The variation in the plasma concentration of the two pro-inflammatory cytokines IL-1β and IL18, between a baseline level measured the day before the operating room (D-1) and 24 hours (D1) after cardiac surgery with ECC. The variation in their concentrations is measured between D-1 and D1 in order to assess the inflammatory response occurring in the first hours post ECC, and mediated by the NLRP3 inflammasome.

SECONDARY OUTCOMES:
Compare the plasma levels of IL-1β and IL18 | Compare between Day-1 and Day 7
  The plasma levels of IL-1β and IL18 will be determined using commercial assay kits (ELISA technique and expressed in pg / mL).

OTHER OUTCOMES:
Compare the plasma concentration of mitochondrial (damage-associated molecular patterns) DAMPS | Compare between Day-1 and Day 7
  Plasma mitochondrial DNA plasma concentration will be achieved by the real-time polymerase chain reaction (PCR). The results will be expressed in number of copies of DNA per microliter.
Compare the level of activation of the NLRP3 inflammasome in circulating blood monocytes | Compare between Day-1 and Day 7
  The level of activation of the NLRP3 inflammasome in circulating blood monocytes, expressed by the number of copies of NLRP3 mRNA measured in quantitative RT-PCR (RT-qPCR) in monocytes isolated from circulating blood.
Compare the plasma concentration of reactive protein C (CRP) the level of activation of the NLRP3 inflammasome in circulating blood monocytes. | Compare between Day-1 and Day 7
  CRP is a protein synthesized by the liver whose expression increases during the acute phase of inflammation

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Martinique, Fort-de-France, Martinique

IPD SHARING:
Plan to Share IPD: No